CLINICAL TRIAL: NCT02136173
Title: Study of Weight Loss Effect of the Sequential Balloons
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, MOHAMED ABDELLATIF, PHD, Mansoura University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sequential balloons
Record Dates: First submitted 2014-05-07; First posted 2014-05-12 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Weight Loss; Balloon
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- sequential balloons (Experimental): effect of weight loss by applying sequential balloons
  Interventions: Device: Heliosphere bag (air filled balloon)

INTERVENTIONS:
Device: Heliosphere bag (air filled balloon) — sequential balloons . Heliosphere bag (air filled balloon)

SUMMARY:
The effect of the balloon on weight loss is investigated by multiple studies. However, the effect of the sequential balloons is not studied yet.

DETAILED DESCRIPTION:
We are aiming to study the effect of the sequential balloons in the patients who had weight loss with the first balloon and they need subsequent balloons to have more weight loss after their first balloons are removed after 6 months.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 45 and weight >120 Kg
* Patients refused to have bariatric surgery.

Exclusion Criteria:

* Esophageal or gastric or duodenal lesions.
* Bleeding disorders.
* uncooperative patients.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2012-12; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
weight loss | 12 months
  study the weight loss in form of KG and BMI before balloon, 6 months after and 12 months after

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Egypt